CLINICAL TRIAL: NCT07116785
Title: A Prospective Double Blind Randomized Controlled Trial to Evaluate the Efficacy and Durability of Accelerated BrainsWay Deep Transcranial Magnetic Stimulation (Deep TMS) Protocol in Obsessive-Compulsive Subjects
Brief Title: Accelerated Rotational Field Deep TMS for Treating OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: Brainsway (Industry)
Responsible Party: Principal Investigator, Dor Shukrun, PhD Student, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0140-22-SOR; 0140-22-SOR (Registry Identifier: Soroka University Medical Center Institutional Registry)
Record Dates: First submitted 2025-08-07; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Deep TMS; Rotational Field
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel assignment, randomized controlled trial comparing the effects of accelerated rotational-field deep transcranial magnetic stimulation versus sham stimulation in patients with OCD
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TMS (Experimental)
  Interventions: Device: BrainsWay Deep TMS HAC/H7-Coil
- Sham TMS (Sham Comparator)
  Interventions: Device: BrainsWay Deep TMS Sham Coil

INTERVENTIONS:
Device: BrainsWay Deep TMS HAC/H7-Coil — Rotational field TMS (rfTMS) is a novel technology where two orthogonal coils are operated with a 90 phase shift between them. The combined electric field vector of rfTMS from both coils rotates up to a complete cycle during the TMS pulse. This method overcomes the inherent limitation of conventional unidirectional TMS by influencing neurons in various orientations (Roth et al., 2020b). This unique advance bears enormous potential for therapeutic applications in various neuropsychiatric disorders. The coil Array includes the H7 coil as the lower coil, and an upper coil perpendicular to it. Hence, the HAC/H7 coil Array induces similar electric field distribution and affects the same brain structures as the H7 coil, but stimulates neurons in various orientations within these regions.
  Arms: Active TMS
Device: BrainsWay Deep TMS Sham Coil — Participants assigned to this intervention will receive sham stimulation using a BrainsWay Deep TMS sham coil that mimics the sensation and acoustic properties of active stimulation but does not deliver effective magnetic pulses to the brain. This condition is used as a placebo control to blind participants and investigators.
  Arms: Sham TMS

SUMMARY:
A Prospective Double Blind Randomized Controlled Trial to Evaluate the Efficacy and Durability of the BrainsWay Rotational Field Deep Transcranial Magnetic Stimulation (Deep TMS) in Obsessive-Compulsive Subjects

DETAILED DESCRIPTION:
This study is a randomized, double-blind clinical trial designed to compare the efficacy of active rfTMS coil targeting the mPFC and ACC with an inactive sham treatment. Conducted over a 13-week period, the trial includes 39 treatment sessions following an accelerated protocol. Eligible participants are randomly assigned in a 1:1 ratio to either the active treatment or sham group. Each daily treatment comprises three sessions separated by 1-hour intervals, resulting in a total treatment duration of 2.5 hours per day. The treatment regimen is structured into three distinct phases (Figure 1): (1) an acute phase (week 1), in which participants are treated for five consecutive days (totaling 15 sessions); (2) a maintenance phase (weeks 2-6), during which participants are treated once per week for five weeks (totaling 15 sessions); and (3) a follow-up phase during which participants are treated every visit at weeks 8, 10, and 13 (totaling 9 sessions). Imaging sessions are conducted at baseline and at the end of the maintenance session.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Diagnosed as suffering from OCD according to the DSM-V.
* Subjects with a YBOCS score of >20.
* If on SRI, patient must be maintained on current dosages (with or without additional antidepressant or psychotropic augmentation for treatment of OCD), at a stable therapeutic dosage for at least 2 months prior to study entry and for the duration of the trial.
* If in CBT, must be in the maintenance stage (i.e., not receiving active training in exposure and response prevention, which is the core component of this treatment). CBT can be with teletherapy but must be for a minimum of ten sessions with a symptom checklist, hierarchy, with exposure and response prevention therapy.
* Have negative or justified responses by the investigator to all questions listed on the Transcranial Magnetic Stimulation Safety Screening questionnaire (TASS).
* According to the treating physician the subject is compliant with taking medication, if applicable.
* Subject is capable and willing to provide informed consent and assent.
* Willing and able to adhere to the treatment schedule.
* All comorbid diagnoses have been stable for 3 months and anticipated to be stable for the 3 months treatment duration.

Exclusion Criteria:

* Subjects diagnosed as suffering from any other Axis I diagnosis as the primary diagnosis.
* Comorbid, secondary psychiatric diagnoses are unstable and are likely to require changes in therapeutic regimens even if OCD improves.
* Present suicidal risk as assessed by the investigator using the Columbia Suicide Severity Rating Scale, brief mental status exam and psychiatric interview or a history of attempted suicide in the past year.
* History of epilepsy or seizure (EXCEPT those therapeutically induced by ECT and febrile seizures in infancy).
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure, or history of significant head trauma with loss of consciousness for greater than or equal to 5 minutes.
* History of head injury necessitating cranial surgery or prolonged coma.
* History of any ferromagnetic of conductive material in the head including the eyes and ears (outside the mouth).
* Known history of any metallic particles in the eye, implanted neurostimulators, intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes).
* History of significant hearing loss.
* Subjects with significant neurological disorder or insult
* Substance use disorder within the past 6 months (except nicotine and caffeine and based on the doctor's judgment).
* Currently participating in another therapeutic clinical study.
* Suffer from an unstable physical, systemic and metabolic disorder such as unstable blood pressure, unstable blood sugar, or acute, unstable cardiac disease.
* Subject on high doses of antidepressant or psychotropic medications, which are known to lower the seizure threshold. Subject is currently on Clomipramine.
* Significant possibility of death within eighteen months of baseline.
* Planned surgeries that will interrupt the study schedule within four months of baseline.
* Women who are breast-feeding.
* Women who are pregnant or with suspected pregnancy.
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2027-06-14 (Estimated); Study Completion 2028-12-14 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (YBOCS) | 6 weeks
  Change in YBOCS scores from baseline to the end of six weeks between the active Deep TMS and Sham treatment groups.
  Scores on the YBOCS range from 0 (no Symptoms) to 40 (Extreme Symptoms).

SECONDARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (YBOCS) | 13 weeks
  Change in YBOCS scores from baseline to the end of thirteen weeks between the active Deep TMS and Sham treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Zangen, Prof., Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: Undecided